CLINICAL TRIAL: NCT01574794
Title: Changes in Running Gait Biomechanics Following an Intervention Program in Older Runners
Brief Title: Exercise Intervention and Running Biomechanics in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Running Injury Clinic (Other); Alberta Heritage Foundation for Medical Research (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Reginaldo Fukuchi, MSc, MSc, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIC-CAPES-001
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Aging; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strengthening Exercises (Experimental): Recreational older runners recruited from local community
  Interventions: Other: Muscle strengthening exercises
- Stretching Exercises (Experimental): Recreational older runners recruited from local community
  Interventions: Other: Muscle stretching exercise
- Control Group (No Intervention): Recreational older runners recruited from local community

INTERVENTIONS:
Other: Muscle strengthening exercises — The group will perform 8-week home based muscle strengthening exercises with 8 weekly supervised sessions which will be conducted by a rehabilitation specialist.
  Arms: Strengthening Exercises
Other: Muscle stretching exercise — The group will perform 8 week home based exercise intervention with 8 weekly supervised sessions which will be conducted by a rehabilitation specialist
  Arms: Stretching Exercises

SUMMARY:
The goal of this study is to understand the effects of muscle strengthening and stretching exercise intervention on isometric muscle strength, joint flexibility and running biomechanical patterns in older recreational runners. To do so, the subjects will be assessed before and after they engage in a 8-week exercise intervention program.

ELIGIBILITY:
Inclusion Criteria:

* no injuries of the lower extremity within 3 months prior to participation
* running recreationally 2-3 times/week
* familiar and comfortable with treadmill running
* in good health upon entry into the study
* no use of orthotics in the shoe

Exclusion Criteria:

* lower extremity injury within the last 3 months
* surgery to the lower extremity within the last 8 months
* head injury/vestibular disorder within the last 6 months
* inability to speak or read English.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of biomechanical movement patterns | 8 weeks
  Biomechanical measurements (kinematics and kinetics) will be taken at baseline and at 8 weeks of intervention.

SECONDARY OUTCOMES:
Changes in isometric muscle strength and joint flexibility | 8 weeks
  Measurements of isometric muscle strength and joint flexibility will be taken at baseline and at 8 weeks of intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Reed Ferber, PhD, Principal Investigator — Running Injury Clinic, Faculty of Kinesiology, University of Calgary
Locations (1):
- Running Injury Clinic, Calgary, Alberta, Canada